CLINICAL TRIAL: NCT04102839
Title: PWS Outcome Assessment Study
Brief Title: PWS Outcomes Assessment Study
Status: Completed | Type: Observational
Sponsor: Soleno Therapeutics, Inc. (Industry)
Collaborators: Casimir Trials (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAS-SOL001-01
Record Dates: First submitted 2019-08-23; First posted 2019-09-25 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; PWS
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Qualitative Interview

SUMMARY:
This is a longitudinal study during which qualitative interviews will be conducted with caregivers of Soleno C601/C602 study subjects. There is an additional option for caregivers to collect video data of PWS patients doing specific activities of daily life.

The purpose of this study is to understand the real-world and nuanced impact of a potential therapeutic on individual PWS patients. The results of this study will complement the outcomes being captured during the Soleno C601/C602 clinical studies.

There is no treatment or intervention associated with this study.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria for Interviews:

Eligible caregivers must:

* Be willing and able to provide informed consent in English
* Care for a C601/C602 trial subject or potential trial subject
* Have access to a smartphone or the internet
* Be able to converse in English

Key Inclusion Criteria for Video Capture:

Eligible PWS participants for the optional daily life video capture must:

* Be willing and able to provide informed consent or assent.
* Be enrolled in the C601/C602 trial
* Be able to converse in English
* Have a caregiver who has access to an Apple or Android smartphone or has internet access and is willing to use a wi-fi-only device to record and upload videos
* Have a caregiver who is willing and able to record activity videos

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of PWS patients who are participating in Soleno C601 and C602 Clinical Studies.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Meaningful Change in Symptom Categories | From baseline for interview #2 (Week 13-16), From baseline for interview #3 (Week 26-28), From baseline for interview #4 (Week 65-67)
  The percentage of caregivers reporting meaningful change in each of the symptom categories in the Study C601 treated arm versus the Study C601 placebo arm as measured by the five-point quantification scale anchored in the qualitative questions (Scale: 1=very meaningful negative change, 2=slightly meaningful negative change, 3=no meaningful change, 4=slightly meaningful change, 5=very meaningful positive change)

CONTACTS AND LOCATIONS:
Locations (1):
- Casimir Trials, Plymouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No